CLINICAL TRIAL: NCT03146091
Title: Study on Outpatient Treatment of Uncomplicated Diverticulitis With Either Antibiotic or Nonantibiotic Treatment: a Randomized Pilot Trial
Brief Title: Outpatient Treatment of Uncomplicated Diverticulitis With Either Antibiotic or Nonantibiotic Treatment
Acronym: MUD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Dr. Marylise Boutros, Colorectal Surgery Attending Staff, Assistant Professor of Surgery at McGill University, Jewish General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CODIM-MBM-17-020
Record Dates: First submitted 2017-04-18; First posted 2017-05-09 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Uncomplicated Diverticular Disease
Keywords: Antibiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Outpatient nonantibiotic treatment (Experimental)
  Interventions: Other: Nonantibiotic treatment of uncomplicated diverticulitis
- Outpatient antibiotic treatment (Active Comparator)
  Interventions: Other: Antibiotic treatment of uncomplicated diverticulitis

INTERVENTIONS:
Other: Nonantibiotic treatment of uncomplicated diverticulitis — Patients randomized to this arm will be treated without antibiotics in the outpatient setting. Pain will be managed with appropriate analgesia as per protocol.
  Arms: Outpatient nonantibiotic treatment
Other: Antibiotic treatment of uncomplicated diverticulitis — Patients randomized to this arm will be treated with antibiotics in the outpatient setting. Pain will be managed with appropriate analgesia as per protocol.
  Arms: Outpatient antibiotic treatment

SUMMARY:
Uncomplicated sigmoid diverticulitis is a common disease in Western countries. Traditional management includes inpatient administration of either oral or intravenous antibiotics with resumption of oral intake as symptoms improve. Recent literature has however questioned both inpatient and antibiotic treatment. Indeed, both inpatient and antibiotic treatment are associated with non-negligible risks to patients. The aim of this trial is to assess the feasibility of a randomized controlled trial designed to determine whether nonantibiotic treatment of uncomplicated diverticulitis is safe in the outpatient setting.

DETAILED DESCRIPTION:
Uncomplicated sigmoid diverticulitis is a common disease in Western countries. Traditional management includes inpatient administration of either oral or intravenous antibiotics with resumption of oral intake as symptoms improve. Recent literature has however questioned both inpatient and antibiotic treatment. Indeed, both inpatient and antibiotic treatment are associated with non-negligible risks to patients. The aim of this trial is to assess the feasibility of a randomized controlled trial designed to determine whether nonantibiotic treatment of uncomplicated diverticulitis is safe in the outpatient setting. It is designed as a pilot non-inferiority blinded randomized controlled trial. The estimated length of this pilot trial is 1 year. The target population is capable adults of who have a CT-diagnosed episode of uncomplicated diverticulitis who present to the Jewish General Hospital Emergency room.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 and < 90 years old
2. Capable of giving informed consent
3. Lower abdominal pain and/or tenderness
4. Confirmed affection of left colon, including descending and sigmoid colon
5. Confirmed episode of acute uncomplicated diverticulitis on computed tomography (CT) scan defined as wall edema with or without fat stranding. Limited pericolic air with bubbles less than 5 mm in size, and less than 5cm from the colon wall, will be included as uncomplicated diverticulitis. Scan must be performed prior to enrollment and assessment for illegibility. The initial scan is not a study-specific procedure.

Exclusion Criteria:

1. CT scan shows complicated diverticulitis as defined by the presence of intraperitoneal free perforation (i.e. intraperitoneal contrast extravasation if intra-rectal contrast given, free air under diaphragms, disseminated intraperitoneal air), abscess, obstruction, fistulisation, and phlegmon.
2. Suspicion of colorectal cancer on CT scan
3. Immunosuppression (including but not exclusively insulin-dependent diabetes mellitus, chronic liver disease, ongoing chemotherapy, chronic renal failure with hemodialysis, corticosteroid and immunosuppressive medication)
4. Pregnancy and breastfeeding
5. Any comorbid infection requiring
6. High fever (≥ 38.5 ºC)
7. Significant leukocytosis (> 15 g/dL)
8. Abdominal pain worsening in the emergency, impeding ambulation and/or eating
9. Evidence of generalized peritonitis on physical exam
10. Intolerance to oral intake and/or persistent vomiting
11. Marked abdominal distension and/or signs of ileus on CT scan
12. Noncompliance/unreliability for return visits/lack of support system
13. Failed outpatient treatment not previously included in study within last 30 days
14. Cognitive, social or psychiatric impairment
15. For patients aged 65 years or older, a Charlson Comorbidity Score ≥ 5 as calculated on the following website: https://www.thecalculator.co/health/Charlson-Comorbidity-Index-(CCI)-Calculator-765.html 19-20.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2017-05-20 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Participants' retention rate as assessed by the number of participants retained in the study from screening to the end of follow-up. | 1 year
  The primary outcome pertains to the feasibility of a non-inferiority randomized controlled trial. The study group's main concern is that accrual will be impeded by the important change in clinical management that nonantibiotic treatment of uncomplicated diverticulitis requires. Also, the study group is concerned that patients may be lost to follow-up. For these reasons, the primary outcome is the retention rate of patients from screening to the end of follow-up. The rate will be calculated according to (1) the proportion of participants screened but not randomized, and (2) the proportion of participants lost to follow-up.

SECONDARY OUTCOMES:
Treatment failure | 1 year
  Treatment failure is defined as persistence, increase or recurrence of abdominal pain and/or fever, inflammatory bowel obstruction, need for radiological abscess drainage or immediate surgery due to complicated diverticulitis, need for hospital admission, and mortality during the first 60 days after discharge.

CONTACTS AND LOCATIONS:
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No